CLINICAL TRIAL: NCT01351129
Title: A Phase 1, Single-Dose, Open-Label, Crossover Study To Estimate The Relative Bioavailability Of Two Controlled-Release Formulations Vs. An Immediate Release Formulation Of PF-04991532 In Healthy Adult Subjects
Brief Title: Single Dose Study To Compare Pharmacokinietics Of 3 Different Formulations Of PF-04991532 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B2611009
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Healthy
Keywords: formulation comparison
MeSH Terms: interventions — Akacid-medical-formulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Formulation 1 (Experimental)
  Interventions: Drug: Formulation 1
- Formulation 2 (Experimental)
  Interventions: Drug: Formulation 2
- Formulation 3 (Experimental)
  Interventions: Drug: Formulation 3

INTERVENTIONS:
Drug: Formulation 1 — 150-mg immediate release tablet (single dose)
  Arms: Formulation 1
Drug: Formulation 2 — 150-mg modified release capsule, short duration (single dose)
  Arms: Formulation 2
Drug: Formulation 3 — 150-mg modified release capsule, long duration (single dose)
  Arms: Formulation 3

SUMMARY:
The primary purpose of this study is to evaluate the pharmacokinetics, safety and tolerability three different formulations of PF-04991532 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (non-childbearing potential) subjects between the ages of 21 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at Screening.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time profile (AUC) | predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12,24,36,48 hrs postdose

SECONDARY OUTCOMES:
Max observed plasma concentration (Cmax) | predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12,24,36,48 hrs postdose
Time of Cmax (Tmax) | predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12,24,36,48 hrs postdose
Concentration at 24 hours postdose (C24hr) | 24 hrs postdose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2611009&StudyName=Single%20Dose%20Study%20To%20Compare%20Pharmacokinietics%20Of%203%20Different%20Formulations%20Of%20PF-04991532%20In%20Healthy%20Volunteers